CLINICAL TRIAL: NCT02856789
Title: Determination of Fibrin Activity in Plasma on STA-R® Prototype
Acronym: FAST
Status: Completed | Type: Observational
Sponsor: Diagnostica Stago R&D (Industry)
Collaborators: Hôpital d'Instruction des armées Percy (Unknown)
Responsible Party: Sponsor
Other Study IDs: FAST STUDY 2016-A00869-42
Record Dates: First submitted 2016-07-08; First posted 2016-08-05 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Blood Coagulation Disorders; Thrombotic Disorders; Hemorrhagic Disorders; Trauma
Keywords: Fibrin structure; Coag-Lysis assay; Fibrin formation; Fibrinolysis; TEG 5000; TEG 6S; Coagulo-lytic balance; Normal range; Thromboelastography
MeSH Terms: conditions — Blood Coagulation Disorders; Hemorrhagic Disorders; Wounds and Injuries | interventions — Thrombelastography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fresh and frozen citrated Poor Platelets Plasma 200 Healthy volunters 50 Patients without coagulation disorder 650 Patients with coagulation disorder
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy volunteers (HV): HV without any known treatment, without any coagulation trouble and with normal hemostasis results.
  FS and TEG will be processed to define the most relevant parameters for normal range and the correlation between both assays.
  Tests performed on HV :
  * Routine hemostasis tests
  * Fibrin structure (FS)
  * Thromboelastography (TEG)
  * Specialized hemostasis tests
  Interventions: Other: Routine hemostasis tests; Other: Fibrin structure (FS); Other: Thromboelastography (TEG); Other: Specialized hemostasis tests
- Patients without coagulation disorder: Hospitalized patients without coagulation disorder or abnormal hemostasis and hematological results and witout ongoing treatment (mainly anticoagulant treatment). FS and TEG will be processed to determine the most relevant parameters to discriminate patients from normal range and the correlation between assays.
  Tests performed on patients :
  * Routine hemostasis tests
  * Fibrin structure (FS)
  * Thromboelastography (TEG)
  Interventions: Other: Routine hemostasis tests; Other: Fibrin structure (FS); Other: Thromboelastography (TEG)
- Patients with coagulation disorders: Hospitalized patients with coagulation disorders, mainly trauma patients or abnormal hemostasis and hematological results, mainly decreased fibrinogen level . FS and TEG will be processed to determine the most relevant parameters to discriminate patients from normal range and the correlation between assays.
  Tests performed on patients :
  * Routine hemostasis tests
  * Fibrin structure (FS)
  * Thromboelastography (TEG)
  Interventions: Other: Routine hemostasis tests; Other: Fibrin structure (FS); Other: Thromboelastography (TEG)

INTERVENTIONS:
Other: Routine hemostasis tests — Prothrombin Time (PT),Thrombin Time (TT), Activated Partial Thromboplastin Time (APTT), Fibrinogen, D-Dimers
Other: Fibrin structure (FS) — FS will be determined on STA-R® prototype at Percy and at Stago
Other: Thromboelastography (TEG) — Thromboelastography will be processed on TEG® at Percy
Other: Specialized hemostasis tests — Coagulation factors
  Groups: Healthy volunteers (HV)

SUMMARY:
The purpose of the study is to give the proof of concept of the Fibrin structure assay on STA-R® prototype. It aims to identify the parameters which discriminate the pathologic from the normal population. Secondary objectives are to determine the precision of the assay, to record the Fibrin activity, comparatively with thromboelastography on TEG®, in a coagulation activation assay and in a coagulation-lysis assay.

DETAILED DESCRIPTION:
Background. Fibers thickness of the fibrin clot plays an important role on the clot stability and its resistance to the fibrinolysis. The innovative concept, based on the relationship between light spectrum through the fibrin clot and its fiber nanostructure (C.Dassi et al, ISTH 15ABS-3593), thanks to a multi-wavelength STA-R® prototype, was simplified by using a coag-lysis assay (An international study on the feasibility of a standardized combined plasma clot turbidity and lysis assay: SSC communication ; Pieters et al. ; JTH 2018) Preliminary results suggest that this new automated FS method provides new data on clot analysis and could be a useful tool in clinical practice in the management of hemostasis disorders. This study is extended to begining of march 2019.

Main objective. This study aims to determine the precision, the normal range of the FS method in comparison with Thromboelastography on TEG® and discriminate patients from healthy volunteers (HV).

Recruitment. 200 healthy volunteers without any known coagulation troubles, enrolled during coagulation testing or blood donation.

50 hospitalized patients or patients from consultations, without ongoing treatment (particularly anticoagulant treatment), with a normal hemostasis screening (Prothombin Time, Activated Partial Prothombine Time and Fibrinogen Level).

650 hospitalized patients for any pathology known and able to induce a increase or a decrease of the fibrinogen level, mainly from trauma patients and enrolled during coagulation testing.

The study is conducted in compliance with French regulation after ethics approval.

FS Assays. The FS determinations on STA-R® prototype and those on TEG® will be realized with fresh plasmas and whole blood samples respectively at the Hôpital d'Instruction des armées Percy. The screening tests (PT, APTT, and Fibrinogen) on STA-R® Evolution and the measurement of FS on a second STA-R® prototype will be performed with frozen plasmas at STAGO laboratory.

Statistical analysis of results. A statistical analysis will determine the most relevant parameters in the discrimination of the pathologic population from the normal population, and the quality control precision. Then, statistical analysis will compare STA-R® prototype method to the TEG® method to point out the most populations discriminating method.

ELIGIBILITY:
Inclusion Criteria:

* Patients and healthy volunteers with non-opposition to participate in the evaluation
* Healthy volunteers : from 18 years to 70 years
* Patients : minimum age limit 18 years - no maximum age limit

Exclusion Criteria:

* Healthy volonteers with ongoing treatment
* Healthy volonteers with abnormal hemostasis results

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volonteers from Centre de Transfusion des Armées (CTSA) and from Centre Principal d'Expertise Médicale du Personnel Navigant (CPEMPN).
  Percy hospital patients from at least: Emergency Unit (EU), Intensive Care Unit (ICU), Burnt Treatment Center (BTC), Hematology department.
Sampling Method: Non-Probability Sample
Enrollment: 913 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Dynamic evolution of the number of protofibrils | 12 months
  Evolution of the Fibrin structure (FS) measurement will be performed on two plasma groups, the first group is constituted with fresh healthy volunteers and the second one with fresh patients. Coagulolytic balance will be measured with FS method. In addition, a normal range will be determined on fresh healthy volunteers without any known coagulation troubles. Fibrin structure is processed to determine the most relevant parameters to discriminate patients from normal range and the correlation between assays.
Dynamic evolution of fibrin formation | 12 months
  Evolution of the optical density measurement and calculating the fibrinogen level and coagulolytic balance

SECONDARY OUTCOMES:
Thromboelastography measurement on TEG 5000 | 12 months
  Thromboelastography will be performed on two plasma groups, the first group is constituted with fresh healthy volunteers and the second one with fresh patients. Viscoelastic clot parameters will be determined on TEG 5000. Thromboelastography is processed to determine the most relevant parameters to discriminate patients from normal range and the correlation between assays.
Prothrombin Time (PT) | 12 months
  These assays will be performed at Stago on all samples from healthy volunteers (HV) and patients to allow the biological confirmation of normal samples from HV group. In case of one abnormal result, the sample is considered as not relevant for the normal range determination of Fibrin Structure measurement and will be discarded from HV group.
Thrombin Time (TT) | 12 months
  These assays will be performed at Stago on all samples from healthy volunteers (HV) and patients to allow the biological confirmation of normal samples from HV group. In case of one abnormal result, the sample is considered as not relevant for the normal range determination of Fibrin Structure measurement and will be discarded from HV group.
Activated Partial Thromboplastin Time (APTT) | 12 months
  These assays will be performed at Stago on all samples from healthy volunteers (HV) and patients to allow the biological confirmation of normal samples from HV group. In case of one abnormal result, the sample is considered as not relevant for the normal range determination of Fibrin Structure measurement and will be discarded from HV group.
Fibrinogen | 12 months
  These assays will be performed at Stago on all samples from healthy volunteers (HV) and patients to allow the biological confirmation of normal samples from HV group. In case of one abnormal result, the sample is considered as not relevant for the normal range determination of Fibrin Structure measurement and will be discarded from HV group.
D-Dimers | 12 months
  These assays will be performed at Stago on all samples from healthy volunteers (HV) and patients to allow the biological confirmation of normal samples from HV group. In case of one abnormal result, the sample is considered as not relevant for the normal range determination of Fibrin Structure measurement and will be discarded from HV group.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Foissaud, M D, Principal Investigator — Hôpital d'Instruction des armées Percy; Geneviève Contant, Ph D, Study Director — Diagnostica Stago SAS
Locations (1):
- Hôpital d'Instruction des armées Percy - Laboratoire d'Hématologie, Clamart, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yeromonahos C, Polack B, Caton F. Nanostructure of the fibrin clot. Biophys J. 2010 Oct 6;99(7):2018-27. doi: 10.1016/j.bpj.2010.04.059. PMID 20923635
- [Background] Zabczyk M, Undas A. Plasma fibrin clot structure and thromboembolism: clinical implications. Pol Arch Intern Med. 2017 Dec 22;127(12):873-881. doi: 10.20452/pamw.4165. Epub 2017 Dec 11. PMID 29225327
- [Background] Pieters M, Philippou H, Undas A, de Lange Z, Rijken DC, Mutch NJ; Subcommittee on Factor XIII and Fibrinogen, and the Subcommittee on Fibrinolysis. An international study on the feasibility of a standardized combined plasma clot turbidity and lysis assay: communication from the SSC of the ISTH. J Thromb Haemost. 2018 May;16(5):1007-1012. doi: 10.1111/jth.14002. Epub 2018 Apr 15. No abstract available. PMID 29658191